CLINICAL TRIAL: NCT02223442
Title: Cognitive Study on the Use of Central Analgesic Drugs in the Management of Chronic Pain
Brief Title: Central Analgesic Drugs for the Treatment of Chronic Pain
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Parma (Other)
Responsible Party: Principal Investigator, Christian Compagnone, MD, University of Parma
Other Study IDs: opioids for chronic pain
Record Dates: First submitted 2014-08-20; First posted 2014-08-22 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2012-11

CONDITIONS: Chronic Pain
Keywords: chronic pain; central analgesic drugs; adherence to therapy; side effects; quality of life; MOR-NRI drugs
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Chronic pain is defined as pain that persists after healing of the wound that caused it, and can occur even in the absence of any obvious pathological trigger. In our country, there is a growing interest in the proper management of the disease "pain".

Pain is also the first symptom of the disease in 20 -50% of patients with neoplastic disease and from 75% to 90% of patients with advanced cancer suffers from chronic pain .

However, pain management is mostly inadequate. This study aims to assess the Italian clinical practice in reference to the pharmacological management of chronic pain by health professionals involved in the treatment of pain in some centers belonging to the Italian network of pain therapy.

DETAILED DESCRIPTION:
Chronic pain is defined as pain that persists after healing of the wound that caused it, and can occur even in the absence of any obvious pathological trigger. In our country, there is a growing interest in the proper management of the disease "pain".

In fact, the Ministry of Health, first in Europe, introduced a law in 2010 (March 15, 2010, No. 38) to provide for the sick, cancer or not, easy access to the necessary care and to provide specialists a specific training course.

Pain is also the first symptom of the disease in 20 -50% of patients with neoplastic disease and from 75% to 90% of patients with advanced cancer suffers from chronic pain (Marcus 2011).

The "pain disease" is one of the most common causes of access to medical care so it should be recognized as a complex health and research problem, being one of the most expensive and investigated conditions in our society (Pizzo and Clark, 2012; Gupta et al. , 2010; Dagenais et al., 2008).

It has a significant impact on the subjective perception of health status, influence daily activities and is associated with symptoms of depression and other psychological problems that affect the quality of life of the patient (end of 2011 Gureje et al., 1998; Bair et al., 2003, Portenoy, 1996).

However, pain management is mostly inadequate for several medical and social reasons: difficulty in defining the complexity of its pathophysiology, difficulty in finding animal models useful for the development of analgesic drugs, difficulty in finding clinical models predictive of drug efficacy / security, lack of recognition of pain as a health issue and not adequate academic training.

A recent survey in Europe uncovered alarming data: 40% of surveyed patients (46,394) reported an inadequate treatment of accused pain (Breivik et al., 2006).

There are also several open questions regarding the research on the most powerful analgesic drugs used: opioids (Galer et al 1992).

There is no specific experimental model able to solve the three most pressing problems: the predictability of the patient's response, efficacy and safety of opioids.

There is no scientific evidence for the efficacy / safety of long-term use of opioids in chronic pain (Chapman et al., 2010; Manchikanti et al., 2011).

A recent review showed that approximately 22% of patients, suffering from chronic pain and on opioid therapy, suspends therapy for the occurrence of side effects and 5-10% of patients suspend it for a not proper control of pain symptoms (Noble et al., 2010).

This study aims to assess the Italian clinical practice in reference to the pharmacological management of chronic pain by health professionals involved in the treatment of pain in some centers belonging to the Italian network of pain therapy.

ELIGIBILITY:
Inclusion Criteria:

* Males and females over the age of 18 years
* Chronic neuropathic and / or nociceptive and / or mixed pain, whereby clinicians considers necessary to start opioid therapy
* Signed informed consent

Exclusion Criteria:

* Males and females aged under 18 years
* Patients already receiving opioid analgesic drugs or drugs of the class MOR-NRI.
* Taking abuse drugs or alcohol abuse
* Patients with contraindications to the use of central analgesic drugs
* Patients who refuse participation
* Prior cognitive impairment or mental retardation
* Severe immunodeficiency (WBC <4,000)
* Severe renal impairment (serum creatinine > 2g/dl or Creatinine clearance <30 ml / h)
* Hepatic impairment (Cholinesterase <2.000UI or INR> 2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with persistent pain syndromes (chronic pain) followed on an outpatient / DH at some Italian centers of Pain Therapy
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
adherence to therapy | 18 months
  to evaluate the proportion of patients who continues therapy with benefit after one month of enrollment

SECONDARY OUTCOMES:
adherence at 6 months | 18 months
  differences between the central analgesic drugs in the percentage of patients who continue therapy (adherence) at 1 month and 6 months
side effects | 18 months
  difference between the central analgesic drugs in the percentage of patients who develop side effects
quality of life | 18 months
  difference between the central analgesic drugs with regard to the improvement of quality of life reported by the patient

CONTACTS AND LOCATIONS:
Overall Officials: Christian Compagnone, Principal Investigator — University of Parma